CLINICAL TRIAL: NCT03403309
Title: Inosine 5'-Monophosphate to Raise of Serum Uric Acid Level in Patients With Multiple System Atrophy: a Multi-center, Randomized Controlled, Double Blind, Parallel Assigned Clinical Trial (IMPROVE MSA Study)
Brief Title: Inosine 5'-Monophosphate to Raise of Serum Uric Acid Level in Patients With Multiple System Atrophy: a Multi-center, Randomized Controlled, Double Blind, Parallel Assigned Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2017-0990
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Multiple System Atrophy
Keywords: Multiple system atrophy; Uric acid; Inosine 5'-monophosphate; Inosine monophosphate; Inosinic acid
MeSH Terms: conditions — Multiple System Atrophy | interventions — Inosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inosine 5'-monophosphate arm (Experimental): Subjects are treated with inosine 5'-monophosphate to increase serum uric acid level.
  Interventions: Drug: 1) Inosine 5'-monophosphate
- Placebo arm (Placebo Comparator): Subjects are treated with placebo not to increase serum uric acid level.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1) Inosine 5'-monophosphate — 1) Subjects are initiated with 1 tablet (500mg of inosine 5'-monophosphate per one tablet) two times per day, and then titrated up by 1 tablet per every visit up to visit 2, i.e. increased up to 2 tablets two times a day by week 6. A maximum limit of elevated serum uric acid level is 9 mg/dL, so that reducing dose of administration may be considered in case of being way over the top of limited level.
  Arms: Inosine 5'-monophosphate arm
Drug: Placebo — 2) Subjects are initiated with 1 tablet (500mg of placebo tablet with inactive therapeutic effect) two times a day, and then titrated up by 1 tablet per every visit up to visit 2, i.e. increased up to 2 tablets two times a day by week 6. A maximum limit of elevated serum uric acid level is 9 mg/dL.
  Arms: Placebo arm

SUMMARY:
A purpose of the present study is to investigate the capability of serum uric acid elevation, safety, and tolerability of inosine 5'-monophosphate in patients with multiple system atrophy with multicenter, randomized, placebo controlled, parallel assigned design. This may provide the cornerstone for future extended trial in multiple system atrophy, a debilitating disease to date.

DETAILED DESCRIPTION:
Background and objective:

Uric acid (UA) is the end product of purine metabolism in human body, which is converted from the precursor metabolite inosine and finally excreted via route of urine and gastrointestinal tract. A high level of UA, usually ≥ 7.0 mg/dL, may lead to development of gout, nephrolithiasis, or to give detrimental effect to a variety of medical diseases, such as chronic kidney disease, cardiovascular disorders, and diabetes. Meanwhile, UA is the very well-known antioxidant, in which the biological antioxidant act as scavenging free radicals (e.g. peroxynitrite), chelating iron, and preventing peroxidation of lipid. Although there have been two faced aspects on UA, antioxidant versus pro-inflammatory potentials, toward neurodegenerative disorders, converging evidences have been highlighting the effects of potential disease modification so far. Given the certain contribution of oxidative stress to the pathogenesis of various neurodegenerative disorders, a therapeutic attempts to anti-oxidation may be promising and feasible. In observational study, ample evidence has been suggested to be beneficial associations between higher uric acid level and lower the risk of disease, clinical severity and progression in Parkinson's disease, Alzheimer's disease, Huntington's disease, amyotrophic lateral sclerosis, ischemic stroke, and even up to myasthenia gravis across clinical, epidemiological, and radiological studies. In addition, on aspect of interventional study, there have been 4 randomized clinical trials of increasing serum uric acid via administration of inosine so far in multiple sclerosis, stroke, amyotrophic lateral sclerosis, and Parkinson's disease. All of the studies have demonstrated reliable capability of increasing serum uric acid level, and favorable safety and tolerability profile. Currently, a phase II trial in Parkinson's disease demonstrated hopeful view in disease modifying strategy by modulating disease progression rate on the inosine administered group with a dose dependent manner.

In case of multiple system atrophy (MSA), there have been a couple of previous reports including increased serum level of UA in MSA compared to healthy control, and strong correlation in serum uric acid level with either motor or cognitive functions. However, no interventional studies have been undertaken to date at all regarding UA. We aimed to investigate the UA elevating capability, safety, and tolerability of inosine 5'-monophosphate, a precursor of uric acid, in MSA patients with randomized, placebo controlled, and parallel assigned design.

Methods:

All participants are randomized to study drugs, either tablet of placebo or inosine 5'-monophosphate, in 1 to 1 ratio and then undergo scheduled titration. Study drugs are initiated with 1 tablet 2 times per day, and then titrate up by 1 tablet per every visit up to visit 2. That is, 1 tablet two times per day for initial 2 weeks, 1 tablet three times per day from next week 3 to 4, and 2 tablets two times per day from next week 4 to 6, and then maintain throughout to week 24. Laboratory tests including serum uric acid level, urine analysis, and stone analysis are scheduled to be checked at time of week 2, 4, 6, 12, 18, and 24, respectively. A maximum limit of elevated serum uric acid level is 9 mg/dL, and thus reducing dose of administration may be considered in case of exceeding the limited level. Comparison of the extent of altered serum uric acid level, safety, and tolerability from baseline to week 24 will be analyzed after study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who met the clinical criteria of either probable or possible multiple system atrophy, age ranged from 19 to 75 at their onset of symptom.
2. Subjects who underwent brain magnetic resonance imaging or 18F-fluorodeoxyglucose positron emission tomography at the time of their diagnosis in which showed any findings compatible to multiple system atrophy, such as cerebellar or putaminal atrophy, putaminal hyperintense rim or iron accumulation, hot cross bun sign or T2 high signal intensities on middle cerebellar peduncle, and decreased glucose metabolism on putamen or cerebellum.
3. Total score of unified multiple system atrophy rating scale 30 or more at baseline screening.
4. Serum uric acid level ≤ 6.0 mg/dL at baseline screening.

Exclusion Criteria:

1. Prior history of gout, nephrolithiasis, stroke, or chronic kidney disease.
2. Presentation of urine pH ≤ 5.0 or uric acid crystalluria on urine analysis at baseline screening.
3. Subject who showed febrile condition or have any sort of unstable and hopeless disorders.
4. Subjects on following medications undergo 4 weeks of wash-out period, and then not co-administered at all over study duration: co-enzyme Q, creatine, daily vitamin E 50 IU or more, and daily vitamin C 300 mg or more.
5. Presence of psychiatric or cognitive impairment by which interrupt to carry out the whole process of the study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Serum uric acid elevation | Baseline to Week 24
  Serum uric acid elevation is defined as an altered level of serum uric acid from baseline to week 24. A laboratory test is scheduled to be checked at time of week 2, 4, 6, 12, 18, and 24, respectively.
Safety | Baseline to Week 24
  Safety is defined as an occurrence of any adverse events during whole study period.
Tolerability | Baseline to Week 24
  Tolerability is defined as the participants who complete the current study with neither discontinuation nor being unable to increase the study drug for at least 12 weeks or longer due to any adverse event across whole study period.

SECONDARY OUTCOMES:
Unified Multiple System Atrophy Rating Scale (UMSARS) | Baseline and Week 24, respectively
  Altered level of UMSARS from baseline to week 24.
Mini Mental Status Exam (MMSE) | Baseline and Week 24, respectively
  Altered level of MMSE score from baseline to week 24.
Montreal Cognitive Assessment (MoCA) | Baseline and Week 24, respectively
  Altered level of MoCA score from baseline to week 24.
Geriatric Depression Scale (GDS) | Baseline and Week 24, respectively
  Altered level of GDS from baseline to week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Yonsei University College of Medicine, Seoul, Seou, South Korea

IPD SHARING:
Plan to Share IPD: No